CLINICAL TRIAL: NCT02147561
Title: A Safety and Efficacy Study of BOTOX® in Korean Adults With Chronic Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-148
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botulinum toxin Type A (Experimental): Botulinum toxin Type A injected across specific head and neck muscles on Day 0.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A injected across specific head and neck muscles on Day 0.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® treatment in Korean adults with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Ethnically Korean with a diagnosis of chronic migraine

Exclusion Criteria:

* Anticipated need for botulinum toxin treatment for any reason other than chronic migraine during the study
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 280
Completed | 276
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Subjects who didn't receive BOTOX | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included patients enrolled in the study who received study drug. The Safety Population was used to assess the baseline characteristics.
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 279
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.81 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Events
Description: An Adverse Event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: 28 Days
Population: Safety Population: patients enrolled in the study who received study drug
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 279
Percentage of Patients | 24.37

2. Secondary Outcome: Change From Baseline in Headache Impact Test-6 (HIT-6) Total Score
Description: The HIT-6 is a 6 question 5-point scale used to measure the impact of headaches on daily life. The total score ranged from 36 (no impact) to 78 (worst impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Day 28
Population: Efficacy Population: patients enrolled in the study, who received study drug, and who had an efficacy assessment
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 276
Scores on a Scale
  Baseline | 67.54 (5.83)
  Change from Baseline at Day 28 | -7.32 (7.98)

3. Secondary Outcome: Physician Global Assessment of Outcome on a 3-Point Scale
Description: Physicians evaluated patient migraines as improved, no change, or worse compared to baseline.
Time Frame: Baseline, Day 28
Population: Efficacy Population: patients enrolled in the study, who received study drug, and who had an efficacy assessment
Measure: Number; unit: Patients
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 276
Patients
  Improved | 200
  No Change | 72
  Worse | 4

ADVERSE EVENTS:
Description: The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs). The Safety Population included patients enrolled in the study who received study drug.
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 4/279
Other Adverse Events (participants affected / at risk) | 38/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=279)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Migraine (Nervous system disorders) | 1
Common Cold (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=279)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 24
Ptosis (Nervous system disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.